CLINICAL TRIAL: NCT06770647
Title: Predicting Outcomes of Breast-Conserving Surgery in Breast Cancer Patients Using the Modified 5-Item Frailty Index
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2013P001244
Record Dates: First submitted 2024-12-22; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Retrospective Study
Keywords: mFI-5; Modified 5-Item Frailty Index; Breast conserving surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Breast cancer is the most common malignancy among women worldwide, with breast-conserving surgery (BCS) being a key treatment. The modified 5-item frailty index (mFI-5), a well-validated tool for assessing frailty, has shown predictive utility in other surgical contexts but remains under-explored in BCS.

Methods: Using the American College of Surgeons National Surgical Quality Improvement Program database (2008-2021), the investigators identified adult female breast cancer patients who underwent BCS. Frailty was assessed using the mFI-5, scored from 0 to 5, with higher scores indicating greater frailty. Multivariable logistic regression was employed to evaluate associations between mFI-5 scores and postoperative outcomes.

Main question: Can the mFI-5 predict adverse postoperative outcomes in breast-conserving surgery patients?

ELIGIBILITY:
Inclusion Criteria

* Data from 14 annual datasets (2008-2021).
* Female breast cancer patients identified using diagnostic codes:
* ICD-9-CM 174: "Malignant neoplasm of female breast."
* ICD-9-CM 233.0: "Carcinoma in situ of breast."
* ICD-10-CM C50: "Malignant neoplasm of breast."
* ICD-10-CM D05: "Carcinoma in situ of breast."
* Focused on patients diagnosed with breast cancer.
* Further refinement:
* Only patients undergoing breast-conserving surgery (BCS).
* Identified by CPT code 19301: "Partial mastectomy without axillary lymphadenectomy."

Exclusion Criteria

* Missing essential anthropometric data (height and/or weight).
* Implausible BMI values (<7 kg/m² or >250 kg/m², assumed data entry errors).
* Miscoded or vague ICD or CPT entries.
* Concurrent invasive procedures other than BCS.
* Procedures performed by specialties other than general or plastic surgery.
* Male and non-binary patients or those with gender identity disorders (to focus on biologically female cohort).
* Non-elective (emergency) surgical cases.
* Patients with ASA physical status scores >4.
* Patients receiving anesthesia types other than general anesthesia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Study Population: Breast cancer patients with Breast conserving surgery without lymph node removal
Sampling Method: Non-Probability Sample
Enrollment: 96586 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
General data | 30 days
  * Hospital length of stay (in days).
  * Operative time (in minutes).
Any complications | 30 days
  * Patient mortality.
  * (Unplanned) readmission.
  * Surgical and/or medical complications.
Surgical Complications | 30 days
  * Infections (superficial, deep, or organ-space).
  * Wound dehiscence.
  * Bleeding requiring transfusion.
Medical Complications | 30 days
  * Pneumonia.
  * Reintubation.
  * Pulmonary embolism.
  * Ventilator dependence >48 hours.
  * Progressive renal insufficiency.
  * Urinary tract infection.
  * Stroke or cerebrovascular accident.
  * Myocardial infarction.
  * Deep vein thrombosis or thrombophlebitis.
  * Sepsis.
  * Septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana C Panayi, MD PhD, Study Chair — Division of Plastic Surgery, Department of Surgery, Brigham and Women's Hospital, Harvard Medical School, Boston, MA, USA
Locations (1):
- Technische Universität München, Munich, Bavaria, Germany